CLINICAL TRIAL: NCT03758508
Title: Non-invasive Ventilation Versus High Flow Oxygen Through Nasal Cannula in Pneumonia Associated Acute Hypoxemic Respiratory Failure
Brief Title: Non-invasive Ventilation Versus High Flow Oxygen
Acronym: HFO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-022018
Record Dates: First submitted 2018-11-23; First posted 2018-11-29 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Pneumonia-associated Acute Hypoxemic Respiratory Failure
Keywords: Noninvasive ventilation; High flow oxygen nasal cannula; Pneumonia; Acute hypoxemic respiratory failure
MeSH Terms: conditions — Pneumonia; Respiratory Insufficiency | interventions — Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: Efficacy of alternating NIV and HFO compared to HFO alone in the determination of an improvement of PaO2/FiO2 at 21 hours compared to baseline PaO2/FiO2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFO (Active Comparator): Continuous high flow oxygen through nasal cannula for 45 hours; longer if the clinical need persists
  Interventions: Device: High Flow Oxygen nasal cannula
- NIV/HFO (Active Comparator): Alternating noninvasive ventilation (3 hours) and high flow oxygen through nasal cannula (3 hours) for 45 hours; longer if the clinical need persists
  Interventions: Device: High Flow Oxygen nasal cannula; Device: Noninvasive ventilation

INTERVENTIONS:
Device: High Flow Oxygen nasal cannula — High Flow Oxygen nasal cannula
Device: Noninvasive ventilation — In this arm, participants receive noninvasive ventilation through an interface (such as full face mask or oro-nasal mask) alternated with continuous high flow oxygen though humidified nasal cannula
  Arms: NIV/HFO

SUMMARY:
The purpose of the study is to compare the efficacy of alternating Non Invasive Ventilation NIV and High Flow Oxygen HFO compared to High Flow Oxygen HFO alone on gas exchanges and prognosis in pneumonia-associated acute hypoxemic respiratory failure

DETAILED DESCRIPTION:
Both Non Invasive Ventilation (NIV) and High Flow Oxygen through nasal cannula (HFO) are widely used in the setting of hypoxemic respiratory failure of heterogeneous etiology, with no definitive evidence for the superiority of one technique on the other. The purpose of this study is to determine whether alternating NIV and HFO brings any advantage on gas exchanges and prognosis compared to the use of HFO alone in the homogeneous setting of pneumonia-associated acute hypoxemic respiratory failure

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pneumonia based on at least two clinical/laboratory criteria and 1 radiologic criterion among the following:

  * Clinical criteria: fever, cough, purulent sputum, pulmonary examination positive for signs consistent with pneumonia
  * Laboratory criteria: leukocytosis (White blood cells >10000/mcL) or leukopenia (White blood cells < 4000/mcL), rise of the inflammatory markers
  * Radiologic criteria: consolidations at Chest X-ray or CT scan
* Hypoxemic respiratory failure, based on all the following criteria

  * PaO2/FiO2 < 300 after at least 15 minutes conventional oxygen therapy with a FiO2 ≥ 50%
  * Respiratory Rate (RR) ≥ 25/min or need for use of accessory muscles
* Informed consent to study participation

Exclusion Criteria:

* Age < 18 years
* Hypercapnic respiratory failure (pCO2 > 60 mmHg at presentation) such as in Chronic Obstructive Pulmonary Disease
* Presence of another cause of hypoxemic respiratory failure - e.g. pulmonary embolism, acute respiratory distress syndrome (ARDS), pulmonary oedema
* Hemodynamic instability with necessity for use of inotropes and/or vasopressors
* Indication for endotracheal intubation (ETI): Glasgow Coma Scale (GCS) <8, agitation, device intolerance, respiratory arrest
* Immunosuppression (chronic immunosuppressive therapy, clinical history positive for any immunodeficiency - congenital or acquired)
* Do Not Resuscitate (DNR) and Do Not Intubate (DNI) indication
* Tracheostomy
* Nocturnal CPAP ventilation therapy
* Any other condition which the clinician would considered an adjunctive risk for taking part in the study or that would not permit the participant to complete it

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
PaO2/FiO2 improvement | at baseline and at 21 hours
  Efficacy of alternating NIV and HFO compared to HFO alone in the determination of an improvement of PaO2/FiO2 at 21 hours compared to baseline PaO2/FiO2

SECONDARY OUTCOMES:
Intensive Care admission | 30 days
  Rate of admission to Intensive Care Unit in the two arms
Sensation of device comfort and dyspnoea | Baseline, at 21 hours, 45 hours and 30 days after beginning treatment. Optional measures can be taken at 1, 3 and 9 hours
  Evaluation of subjective sensation of device comfort and dyspnoea in the two arms
Time to downgrade to conventional oxygen therapy | 30 days
  Total amount of hours in which the patient needs to be treated with noninvasive ventilation alternate to versus high flow oxygen through nasal cannula
In-hospital mortality | 30 days
  Mortality rate in the 2 arms
New hospital admission | 30 days
  Rate of a new hospital admission within 30 days
PaO2/FiO2 improvement | at baseline and at 45 hours
  Efficacy of alternating NIV and HFO compared to HFO alone in the determination of a change in PaO2/FiO2 at 45 hours compared to baseline PaO2/FiO2
PaO2/FiO2 improvement | at baseline and at 30 days
  Efficacy of alternating NIV and HFO compared to HFO alone in the determination of a change in PaO2/FiO2 at 30 hours compared to baseline PaO2/FiO2

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Grande Ospedale Metropolitano Niguarda, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided